CLINICAL TRIAL: NCT00879086
Title: A Phase II, Multicenter, Randomized, Open-Label Study Comparing Eribulin Mesylate and Ixabepilone in Causing or Exacerbating Neuropathy in Patients With Advanced Breast Cancer
Brief Title: A Study Comparing Eribulin Mesylate and Ixabepilone in Causing or Exacerbating Neuropathy in Participants With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-209
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Oncology
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — eribulin; ixabepilone

ARMS (2):
- Eribulin mesylate (Active Comparator)
  Interventions: Drug: Eribulin Mesylate
- Ixabepilone (Active Comparator)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Eribulin Mesylate — E7389 (eribulin mesylate) given at a dose of 1.4 mg/m^2 as a 2 to 5 minute intravenous (IV) bolus on Days 1 and 8 of a 21-day cycle.
  The Treatment Phase will include six cycles. Patients may enter the Extension Phase for additional cycles following the sixth cycle of treatment.
  Other Names: E7389
  Arms: Eribulin mesylate
Drug: Ixabepilone — Ixabepilone given at a starting dose of 32 or 40 mg/m^2 (as per approved labeling) as a 3-hour IV infusion on Day 1 of a 21-day cycle.
  The Treatment Phase will include six cycles. Patients may enter the Extension Phase for additional cycles following the sixth cycle of treatment.
  Arms: Ixabepilone

SUMMARY:
The purpose of this study in patients with advanced breast cancer is to compare the incidence and severity of neuropathy adverse events for the two treatment groups (eribulin versus ixabepilone) using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 3.0) grading.

ELIGIBILITY:
Inclusion criteria:

1. Female subjects with confirmed locally recurrent or metastatic carcinoma of the breast who have received prior taxane therapy and at least one prior cytotoxic chemotherapy regimen for advanced disease.

Exclusion criteria:

1. Subjects who have received prior ixabepilone therapy.
2. Subjects with prior participation in an eribulin clinical study, even if not assigned to eribulin treatment.
3. Subjects with pre-existing neuropathy Grade greater than or equal to 2.
4. Subjects with a history of diabetes mellitus Type 1 or 2.
5. Subjects with bilateral mastectomy which included bilateral axillary lymph node dissection.
6. Subjects with missing digits required for vibration assessment.
7. Subjects with any other concurrent diseases or conditions that would be expected to interfere with neuropathy assessments, which may include vitamin deficiency, sequelae of cerebrovascular disease, thyroid insufficiency, lumbar or cervical radiculopathy, or alcoholic or inflammatory neuropathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-03-31 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2014-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Northern AZ Hematology and Oncology Associates, Sedona, Arizona
  - Healing Hands Oncology and Medical Care, Hawthorne, California
  - University of Southern California, Los Angeles, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Comprehensive Cancer Care Specialist of Boca, Boca Raton, Florida
  - Robert R. Carroll, MD, PA, Gainesville, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - Medical Specialists of the Palm Beaches, Lake Worth, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Oncology and Hematology Associates of West Broward, Tamarac, Florida
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Heartland Oncology Hematology, Council Bluffs, Iowa
  - Hematology and Oncology Specialists, Marrero, Louisiana
  - Metairie Institute of Comprehensive Health, Metairie, Louisiana
  - Hematology and Oncology Specialists, New Orleans, Louisiana
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Washington County Hospital, Hagerstown, Maryland
  - Josephine Ford Cancer Center, Brownstown, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Health Systems, Detroit, Michigan
  - Henry Ford Medical Center Farmington, West Bloomfield, Michigan
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Joan Knechel Cancer Center, Mount Arlington, New Jersey
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Saint Vincent's Comprehensive Cancer Center, New York, New York
  - Weil Cornell Breast Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Charleston Hematology Oncology Associates PA, Charleston, North Carolina
  - Cancer Center of North Carolina, Raleigh, North Carolina
  - Northwest Cancer Specialists Rose Quarter, Portland, Oregon
  - Northwest Cancer Specialists Hoyt, Portland, Oregon
  - Northwest Cancer Specialists, Tualatin, Oregon
  - Lone Star Oncology, Austin, Texas
  - South Texas Institute of Cancer, Corpus Christi, Texas
  - Northwest Cancer Center, Corpus Christi, Texas
  - Texas Oncology-Sammons Cancer Center, Dallas, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Texas Oncology, PA Bedford, Houston, Texas
  - Texas Oncology, PA, Houston, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Northern Utah Associates, Ogden, Utah
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialist Vancouver, Vancouver, Washington
  - Northwest Cancer Care Specialists, P.C., Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 127 participants were screened. Of these, 104 participants were enrolled and randomized into the study and 23 participants were screen failures (19 failed to meet entrance criteria, 3 failed due to other reason, and 1 failed due to consent withdrawal).
Groups:
- Eribulin Mesylate: Eribulin mesylate was given at a dose of 1.4 milligram per square meter (mg/m^2) as a 2 to 5 minute intravenous (IV) bolus on Days 1 and 8 of a 21-day cycle during the Treatment and Extension Phases. The Treatment Phase included six cycles. Following the sixth cycle of the Treatment Phase, participants who demonstrated clinical benefit could continue treatment during the Extension Phase for an indefinite number of cycles for as long as clinical benefit was sustained (up to 211 weeks).
- Ixabepilone: Ixabepilone was given at a starting dose of 32 or 40 mg/m^2 (as per approved labeling) as a 3-hour IV infusion on Day 1 of a 21-day cycle during the Treatment and Extension Phases. The Treatment Phase included six cycles. Following the sixth cycle of the Treatment Phase, participants who demonstrated clinical benefit could continue treatment during the Extension Phase for an indefinite number of cycles for as long as clinical benefit was sustained (up to 211 weeks).
Period: Overall Study
Arm/Group | Eribulin Mesylate | Ixabepilone
Started | 52 | 52
Safety Analysis Set (SAS) | 51 | 50
Completed | 0 | 0
Not Completed | 52 | 52
Not completed — Adverse Event | 3 | 15
Not completed — Participant choice | 2 | 2
Not completed — Progression of disease | 40 | 26
Not completed — Withdrawal of consent | 2 | 1
Not completed — Other | 4 | 6
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Population: SAS included all randomized participants who received at least one dose of study medication and who had at least one safety assessment following the first dose of study medication.
Groups:
- Eribulin Mesylate: Eribulin mesylate was given at a dose of 1.4 mg/m^2 as a 2 to 5 minute IV bolus on Days 1 and 8 of a 21-day cycle during the Treatment and Extension Phases. The Treatment Phase included six cycles. Following the sixth cycle of the Treatment Phase, participants who demonstrated clinical benefit could continue treatment during the Extension Phase for an indefinite number of cycles for as long as clinical benefit was sustained (up to 211 weeks).
- Total: Total of all reporting groups
Arm/Group | Eribulin Mesylate | Ixabepilone | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (9.83) | 56.9 (10.68) | 54.5 (10.49)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 51 | 50 | 101
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Neuropathy Adverse Events (AEs)
Description: Neuropathy AEs were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 and coded according to the current version of the Medical Dictionary for Regulatory Activities (MedDRA). Neuropathy AEs included the broad list of preferred terms (PTs) defined in the Standard MedDRA Query for Neuropathy and the following additional PTs: neuropathy, hyperesthesia, painful response to normal stimuli, pallanesthesia, and allodynia. If the post-baseline maximum CTCAE grade of the combined term "neuropathy" was greater than the baseline maximum CTCAE grade of the combined term, then the event was considered as treatment emergent neuropathy adverse events per CTCAE grade. For a single participant, 1) a neuropathy AE occurring more than once during the study, whether defined with the same or different MedDRA PTs, was counted only once, 2) a neuropathy AE with different CTCAE grades had only the highest grade AE counted.
Time Frame: From administration of first dose up to approximately 5 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 51 | 50
Percentage of participants | 33.3 [20.8 to 47.9] | 50.0 [35.5 to 64.5]
Statistical Analysis 1: Comparison: Eribulin Mesylate vs Ixabepilone; Test type: Superiority or Other; p = 0.0941, Cochran-Mantel-Haenszel — The two treatment groups were compared, controlling for baseline pre-existing neuropathy (CTCAE Grade 0 or 1) and number of prior chemotherapy regimens (less than or equal to 3 or greater than 3), with both covariates included as binary variables; Difference in proportions = -16.7, 95% CI 2-sided [-36.1 to 2.4] — Extended Mantel-Haenszel test statistics with stratification adjustment for pre-existing baseline neuropathy (CTCAE Grade 0 or 1) and number of prior chemotherapy regimens (greater than or equal to 3 or greater than 3)

2. Secondary Outcome: Percentage of Participants With an Incidence of Treatment-emergent Myalgia/Arthralgia
Description: The incidence rate of TE myalgia/arthralgia was calculated as the percent of participants with TE myalgia/arthralgia. A participant who had an arthralgia or myalgia AE more than once over the course of the study was counted only once in the incidence calculation for myalgia/arthralgia AEs. A participant who had myalgia/arthralgia AEs with different CTCAE grades was counted with the highest CTCAE grade over the course of the evaluation period. If the post-baseline CTCAE grade of the combined term "Myalgia/Arthralgia" was greater than the baseline maximum CTCAE grade of the combined term, the participant had TE myalgia/arthralgia. The 2-sided 95% confidence interval (CI) for incidence rate of TE myalgia/arthralgia was calculated using the Clopper-Pearson method (i.e., the exact method) for each treatment group.
Time Frame: From administration of first dose up to approximately 5 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 51 | 50
Percentage of participants | 19.6 [9.8 to 33.1] | 38.0 [24.7 to 52.8]
Statistical Analysis 1: Comparison: Eribulin Mesylate vs Ixabepilone; Test type: Superiority or Other; p = 0.0492, Cochran-Mantel-Haenszel — Controlled for baseline pre-existing neuropathy (CTCAE Grade 0 or 1) and number of prior chemotherapy regimens (greater than or equal to 3 or greater than 3), with both covariates included as binary variables; Difference in proportions = -18.4, 95% CI 2-sided [-36.0 to -0.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Vibration Perception Threshold (VPT)
Description: The participant-reported questionnaire was used to compare the incidence and severity of neuropathy AEs. Sensory and motor scores were to be analyzed separately using a generalized linear model. Separate subgroup analyses were performed by each stratification variable. VPAT was measured using a Vibratron II device (Physitemp, Inc.) and a modified Two Alternative Forced Choice psychophysical algorithm. VPT was assessed on the ventral surface of the distal index finger (side opposite the nail), contralateral to the side of the mastectomy or primary disease and on the distal fleshy pad of both the right and left great toes (side opposite the nail). If the mastectomy was bilateral, the index finger on the side without axillary lymph node dissection was tested. Data ranged from 0 (invalid) to 20 vu. A lower VPT indicated a greater sensitivity.
Time Frame: Baseline, Treatment Phase: Cycles 2 to 6 (Day 1); Extension Phase: Cycle 9 Day 1, Cycle 12 Day 1, Cycle 15 Day 1 (Each Cycle length=21 days), End of Treatment, Post-treatment Follow-up, Worst Post-baseline result (Up to approximately 5 years)
Population: SAS included all randomized participants who received at least one dose of study medication and who had at least one safety assessment following the first dose of study medication. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: Vibration units (vu)
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 51 | 50
Vibration units (vu)
  Index Finger, Baseline | 1.50 (1.117) | 1.96 (1.373)
  Index Finger, Cycle 2 (Day 1): number analyzed (Participants) | 46 | 42
  Index Finger, Cycle 2 (Day 1) | 0.13 (1.196) | -0.09 (1.641)
  Index Finger, Cycle 3 (Day 1): number analyzed (Participants) | 37 | 29
  Index Finger, Cycle 3 (Day 1) | 0.31 (0.478) | -0.22 (1.762)
  Index Finger, Cycle 4 (Day 1): number analyzed (Participants) | 32 | 25
  Index Finger, Cycle 4 (Day 1) | 0.67 (1.218) | -0.14 (1.588)
  Index Finger, Cycle 5 (Day 1): number analyzed (Participants) | 25 | 20
  Index Finger, Cycle 5 (Day 1) | 0.93 (1.291) | 0.10 (1.828)
  Index Finger, Cycle 6 (Day 1): number analyzed (Participants) | 19 | 18
  Index Finger, Cycle 6 (Day 1) | 1.86 (2.515) | -0.07 (2.213)
  Index Finger, Cycle 9 (Day 1): number analyzed (Participants) | 11 | 12
  Index Finger, Cycle 9 (Day 1) | 1.94 (2.221) | 0.35 (1.144)
  Index Finger, Cycle 12 (Day 1): number analyzed (Participants) | 7 | 2
  Index Finger, Cycle 12 (Day 1) | 0.50 (0.816) | 0.65 (0.354)
  Index Finger, Cycle 15 (Day 1): number analyzed (Participants) | 5 | 1
  Index Finger, Cycle 15 (Day 1) | 0.90 (0.906) | 1.30 (NA) — As only one participant was available here, so standard deviation could not be calculated.
  Index finger, End of Treatment: number analyzed (Participants) | 31 | 34
  Index finger, End of Treatment | 1.23 (2.108) | 0.35 (1.388)
  Index finger, Post-treatment follow-up: number analyzed (Participants) | 5 | 8
  Index finger, Post-treatment follow-up | 1.34 (1.727) | 0.58 (0.991)
  Index finger, Worst post-baseline result: number analyzed (Participants) | 48 | 45
  Index finger, Worst post-baseline result | 1.95 (2.491) | 0.67 (1.721)
  Great toe, Baseline: number analyzed (Participants) | 51 | 49
  Great toe, Baseline | 5.22 (2.393) | 6.60 (3.525)
  Great toe, Cycle 2 (Day 1): number analyzed (Participants) | 46 | 41
  Great toe, Cycle 2 (Day 1) | 0.15 (1.760) | 0.08 (1.988)
  Great toe, Cycle 3 (Day 1): number analyzed (Participants) | 37 | 28
  Great toe, Cycle 3 (Day 1) | 0.49 (2.110) | 0.20 (2.589)
  Great toe, Cycle 4 (Day 1): number analyzed (Participants) | 32 | 24
  Great toe, Cycle 4 (Day 1) | 0.89 (2.037) | 0.82 (3.679)
  Great toe, Cycle 5 (Day 1): number analyzed (Participants) | 26 | 19
  Great toe, Cycle 5 (Day 1) | 1.08 (1.899) | 0.54 (3.645)
  Great toe, Cycle 6 (Day 1): number analyzed (Participants) | 19 | 17
  Great toe, Cycle 6 (Day 1) | 2.28 (2.873) | 0.39 (3.371)
  Great toe, Cycle 9 (Day 1): number analyzed (Participants) | 11 | 12
  Great toe, Cycle 9 (Day 1) | 2.69 (3.711) | 1.34 (2.417)
  Great toe, Cycle 12 (Day 1): number analyzed (Participants) | 7 | 2
  Great toe, Cycle 12 (Day 1) | 1.23 (2.992) | 5.35 (0.636)
  Great toe, Cycle 15 (Day 1): number analyzed (Participants) | 5 | 1
  Great toe, Cycle 15 (Day 1) | 1.12 (3.070) | 3.40
  Great toe, End of treatment: number analyzed (Participants) | 31 | 34
  Great toe, End of treatment | 1.39 (2.208) | 1.71 (2.682)
  Great toe, Post-treatment follow-up: number analyzed (Participants) | 5 | 8
  Great toe, Post-treatment follow-up | 3.34 (2.422) | 1.53 (3.371)
  Great toe, Worst post-baseline results: number analyzed (Participants) | 48 | 44
  Great toe, Worst post-baseline results | 2.39 (2.762) | 2.16 (2.916)

4. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Participant Neurotoxicity Questionnaire (PNQ) Score for Item 1 (Sensory)
Description: The PNQ consisted of 3 parts; Item 1 (sensory) measured numbness, pain, burning or tingling in hands or feet, Item 2 (motor) measured weakness in arms or legs, and Item 3 (activities) measured activities that interfered with daily life. The participant was told that there was no right or wrong answer and their answer should reflect how they currently felt since last completing the PNQ. Sensory scores were analyzed separately. Letter scores (A= none, B=mild, C=moderate, D=moderate to severe, and E=severe) for PNQ were converted to numeric scores A (none)=0, B (mild)=1, C (moderate)=2, D (moderate to severe)=3 and E (severe)=4). Total scores ranged from 0 (minimum severity) to 10 (maximum severity). Higher scores indicated greater severity. Neuropathy AEs that were sensory were evaluated with the PNQ Item 1 (sensory). Categories where no participant showed any shift from baseline to post-baseline for both the arms were not included in the presentation.
Time Frame: Baseline up to approximately 5 years
Population: SAS included all randomized participants who received at least one dose of study medication and who had at least one safety assessment following the first dose of study medication. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 48 | 46
Participants
  A (Baseline) to A (Worst Post-baseline) | 8 | 7
  A (Baseline) to B (Worst Post-baseline) | 9 | 3
  A (Baseline) to C (Worst Post-baseline) | 5 | 4
  A (Baseline) to D (Worst Post-baseline) | 2 | 4
  A (Baseline) to E (Worst Post-baseline) | 0 | 1
  B (Baseline) to A (Worst Post-baseline) | 1 | 1
  B (Baseline) to B (Worst Post-baseline) | 5 | 4
  B (Baseline) to C (Worst Post-baseline) | 2 | 8
  B (Baseline) to D (Worst Post-baseline) | 9 | 5
  B (Baseline) to E (Worst Post-baseline) | 1 | 0
  C (Baseline) to B (Worst Post-baseline) | 0 | 1
  C (Baseline) to C (Worst Post-baseline) | 3 | 4
  C (Baseline) to D (Worst Post-baseline) | 2 | 3
  D (Baseline) to D (Worst Post-baseline) | 1 | 1

5. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Participant Neurotoxicity Questionnaire (PNQ) Score for Item 2 (Motor)
Description: The PNQ consisted of 3 parts; Item 1 (sensory) measured numbness, pain, burning or tingling in hands or feet, Item 2 (motor) measured weakness in arms or legs, and Item 3 (activities) measured activities that interfered with daily life. The participant was told that there was no right or wrong answer and their answer should reflect how they currently felt since last completing the PNQ. Motor scores were analyzed separately. Letter scores (A= none, B=mild, C=moderate, D=moderate to severe, and E=severe) for PNQ were converted to numeric scores A (none)=0, B (mild)=1, C (moderate)=2, D (moderate to severe)=3 and E (severe)=4). Total scores ranged from 0 (minimum severity) to 10 (maximum severity). Higher scores indicated greater severity. Neuropathy AEs that were motor were evaluated with the PNQ Item 2 (motor). Categories where no participant showed any shift from baseline to post-baseline for both the arms were not included in the presentation.
Time Frame: Baseline up to approximately 5 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 48 | 46
Participants
  A (Baseline) to A (Worst Post-baseline) | 8 | 12
  A (Baseline) to B (Worst Post-baseline) | 12 | 3
  A (Baseline) to C (Worst Post-baseline) | 8 | 6
  A (Baseline) to D (Worst Post-baseline) | 2 | 7
  A (Baseline) to E (Worst Post-baseline) | 0 | 1
  B (Baseline) to B (Worst Post-baseline) | 5 | 5
  B (Baseline) to C (Worst Post-baseline) | 4 | 2
  B (Baseline) to D (Worst Post-baseline) | 4 | 4
  C (Baseline) to C (Worst Post-baseline) | 0 | 1
  C (Baseline) to D (Worst Post-baseline) | 0 | 4
  D (Baseline) to A (Worst Post-baseline) | 1 | 0
  D (Baseline) to D (Worst Post-baseline) | 3 | 0
  D (Baseline) to E (Worst Post-baseline) | 1 | 1

6. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline Participant Neurotoxicity Questionnaire (PNQ) Composite Score
Description: The PNQ consisted of 3 parts; Item 1 (sensory) measured numbness, pain, burning or tingling in hands or feet, Item 2 (motor) measured weakness in arms or legs, and Item 3 (activities) measured activities that interfered with daily life. Sensory scores, motor scores and composite scores were analyzed separately. For both item 1 and item 2, letter scores (A=none, B=mild, C=moderate, D=moderate to severe, and E=severe) for PNQ were converted to numeric scores A(none)=0, B(mild)=1, C(moderate)=2, D(moderate to severe)=3 and E (severe)=4. Total scores ranged from 0 (minimum severity) to 10 (maximum severity). Higher scores indicated greater severity. PNQ composite score was defined as the worst of Item 1 and Item 2 score. If neither Item 1 or item 2 score was D or E, but if a box was checked in Item 3, PNQ composite score would be D. Categories where no participant showed any shift from baseline to post-baseline for both the arms were not included in the presentation.
Time Frame: Baseline up to approximately 5 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 48 | 46
Participants
  A (Baseline) to A (Worst Post-baseline) | 3 | 5
  A (Baseline) to B (Worst Post-baseline) | 6 | 1
  A (Baseline) to C (Worst Post-baseline) | 5 | 2
  A (Baseline) to D (Worst Post-baseline) | 2 | 5
  A (Baseline) to E (Worst Post-baseline) | 0 | 1
  B (Baseline) to A (Worst Post-baseline) | 0 | 1
  B (Baseline) to B (Worst Post-baseline) | 5 | 6
  B (Baseline) to C (Worst Post-baseline) | 5 | 6
  B (Baseline) to D (Worst Post-baseline) | 9 | 6
  C (Baseline) to C (Worst Post-baseline) | 2 | 0
  C (Baseline) to D (Worst Post-baseline) | 1 | 3
  D (Baseline) to A (Worst Post-baseline) | 1 | 0
  D (Baseline) to C (Worst Post-baseline) | 0 | 2
  D (Baseline) to D (Worst Post-baseline) | 7 | 7
  D (Baseline) to E (Worst Post-baseline) | 2 | 1

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v.1.0 for target lesions assessed by magnetic resonance imaging and computed tomography and investigator assessment. Participants with unknown or missing responses were treated as non-responders. CR was defined as disappearance of all target lesions. PR was defined as at least a 30 percent (%) decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter. ORR=CR+PR, was presented with 2-sided 95% confidence interval (CI) by the method of Clopper-Pearson method for calculating the exact binomial intervals.
Time Frame: From date of treatment start until disease progression (PD) (Up to approximately 5 years)
Population: Full analysis set (FAS) included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 52 | 52
Percentage of participants | 15.4 [6.9 to 28.1] | 5.8 [1.2 to 15.9]

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization until PD or death due to any cause as determined by the investigator. Disease progression per RECIST v1.0 was defined as at least a 20% relative increase and 5 millimeter absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. The duration of PFS was calculated as the end date minus date of first drug plus 1. For participants who did not have an event (those lost to follow-up or who had not progressed at the date of data cut-off) PFS was censored. The median PFS and corresponding 95% CI was estimated for each treatment group using the Kaplan-Meier method.
Time Frame: From date of treatment start until the date of PD or death from any cause (Up to approximately 5 years)
Population: FAS analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 52 | 52
Days | 104 [80.0 to 129.0] | 95 [73.0 to 186.0]

9. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the number of participants (CR + PR + stable disease (SD) greater than or equal to 6 months) divided by the number of participants in the analysis population. The 95% CI was generated for the clinical benefit rate for each treatment group, and it was based on the Clopper-Pearson method for calculating the exact binomial intervals.
Time Frame: From date of treatment start until PD or death from any cause, whichever occurred first (Up to approximately 5 years)
Population: FAS analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 52 | 52
Percentage of participants | 26.9 [15.6 to 41.0] | 21.2 [11.1 to 34.7]

10. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from first documented CR or PR until PD or death from any cause. It was measured from the time that measurement criteria were met for CR or PR (whichever status was recorded first) until the first date that recurrent or PD was objectively documented. It was defined for participants with a confirmed CR or a confirmed PR. Participants without progressive disease or death were censored. Median duration and 95% CI of the median were estimated for each treatment group, using the Kaplan-Meier method.
Time Frame: From date of first CR or PR until the first documentation of PD or date of death (Up to approximately 5 years)
Population: FAS analysis set included all randomized participants. Number of participants analyzed who had CR or PR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 8 | 3
Days | 169 [60.0 to 246] | NA [NA to NA] — Here, Median and 95% upper and lower CI could not be estimated due to insufficient number of participants with events.

11. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Eribulin and Ixabepilone
Description: General safety was assessed by monitoring all TEAEs and SAEs. TEAEs were reported at a frequency of 0% or greater in the study population.
Time Frame: For each participant, from the first dose till 42 days after the last dose of study treatment (Up to approximately 5 years)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Eribulin Mesylate | Ixabepilone
Number analyzed (Participants) | 51 | 50
Percentage of participants
  TEAEs | 100.0 | 100.0
  SAEs | 37.3 | 34.0

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 42 days after the last dose of study treatment (Up to approximately 5 years)
Description: Treatment-emergent adverse events were reported. All adverse events were graded using National Cancer Institute Common Terminology Criteria (NCI CTCAE) version 3.0. The SAS included all randomized participants who received at least one dose of study medication and who had at least one safety assessment following the first dose of study medication. Of 104 participants randomized into the study, 3 did not receive treatment, 1 in the E7389 Treatment Group and 2 in the Ixabepilone Treatment Group.
Arm/Group | Eribulin Mesylate | Ixabepilone
All-Cause Mortality (participants affected / at risk) | 2/51 | 2/50
Serious Adverse Events (participants affected / at risk) | 19/51 | 17/50
Other Adverse Events (participants affected / at risk) | 51/51 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=51) | Ixabepilone (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia / Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Peripheral Neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=51) | Ixabepilone (N=50)
Neutropenia (Blood and lymphatic system disorders) | 24 | 14
Anaemia (Blood and lymphatic system disorders) | 13 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 7
Leukopenia (Blood and lymphatic system disorders) | 3 | 3
Lacrimation increased (Eye disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 23 | 27
Diarrhoea (Gastrointestinal disorders) | 12 | 12
Vomiting (Gastrointestinal disorders) | 12 | 15
Constipation (Gastrointestinal disorders) | 11 | 10
Dry mouth (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 9
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 19 | 27
Fatigue / Asthenia (General disorders) | 19 | 29
Mucosal inflammation (General disorders) | 11 | 1
Pyrexia (General disorders) | 10 | 5
Chills (General disorders) | 6 | 3
Oedema peripheral (General disorders) | 3 | 5
Asthenia (General disorders) | 2 | 4
Pain (General disorders) | 2 | 4
Chest pain (General disorders) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 2
Pharyngitis (Infections and infestations) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 8 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 0
White blood cell count decreased (Investigations) | 7 | 2
Haemoglobin decreased (Investigations) | 6 | 4
Alanine aminotransferase increased (Investigations) | 5 | 0
Neutrophil count decreased (Investigations) | 5 | 0
Weight decreased (Investigations) | 5 | 0
Platelet count decreased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 17 | 13
Dehydration (Metabolism and nutrition disorders) | 6 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 4
Myalgia / Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 11
Peripheral Neuropathy (Nervous system disorders) | 18 | 23
Neuropathy peripheral (Nervous system disorders) | 16 | 15
Headache (Nervous system disorders) | 7 | 6
Dizziness (Nervous system disorders) | 6 | 4
Dysgeusia (Nervous system disorders) | 4 | 3
Paraesthesia (Nervous system disorders) | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 8
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3
Depression (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other